CLINICAL TRIAL: NCT01016340
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of MCS-5 in Treating Male Oligoasthenospermia (MCS_MOS)
Brief Title: Efficacy and Safety of MCS-5 in Treating Male Oligoasthenospermia
Acronym: MCS_MOS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no safety issues
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCS-5-TWN-a
Record Dates: First submitted 2009-11-17; First posted 2009-11-19 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Male Oligoasthenospermia
Keywords: Male Oligoasthenospermia; MCS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MCS-5 (Active Comparator): Group 1: MCS-5 5 mg/day for 16 weeks;Group 2: MCS-5 10 mg/day for 16 weeks;Group 3: MCS-5 20 mg/day for 16 weeks
  Interventions: Drug: MCS
- Placebo (Placebo Comparator): Group 4: Placebo for 16 weeks
  Interventions: Drug: MCS

INTERVENTIONS:
Drug: MCS — MCS-5 Softgel 5 mg

SUMMARY:
This is a phase II randomized, double-blind, placebo-controlled study where eligible subfertile male subjects (age 20 years).

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects who are 20 years old or older
2. Subjects who are diagnosed as idiopathic oligoasthenospermia
3. Subjects who have a normal baseline hormone profile
4. Subjects who were not able to impregnate female partners in the past 12 months under an active and unprotected sexual life
5. Subject's female partner has no endocrine or genital obstructive disorders and is capable of impregnation.
6. Subjects who have an acceptable baseline liver function
7. Subjects who have a normal baseline renal function.

Exclusion Criteria:

1. Subjects who have been diagnosed as male infertility for more than 5 years.
2. Subjects who have a baseline semen white blood cell count of 1*106/mL.
3. Subjects who have genital/seminal tract obstruction, infection, inflammation or anatomic abnormalities.
4. Subjects whose female partner has been diagnosed as infertility of any kind.
5. Male infertility that is associated with hormonal deficiency/imbalance, poor nutrition, congenital/chromosomal disorders, erectile dysfunction, or psychological disorders.
6. Subjects who plan to undergo artificial insemination of any kind within the study period.
7. Subjects who have been treated with chemotherapy, pelvic irradiation or major pelvic surgery
8. Subjects who will undergo any invasive procedures within the study period
9. Subjects who will undergo any chemotherapy or radiotherapy of any kind during the study period.
10. Subjects who can not or are not willing to undergo the two-week wash-out period for any reasons.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To compare changes in total motile sperm (TMS) between groups from baseline to 16 weeks after treatment | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan